CLINICAL TRIAL: NCT01153282
Title: Physical Functional Side Effects of Taxane Chemotherapy for Breast Cancer
Status: Completed | Type: Observational
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: UPCC 14110
Record Dates: First submitted 2010-06-28; First posted 2010-06-30 (Estimated); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Breast Cancer
Keywords: Breast Cancer patients
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Determine the characteristics of symptoms and functional impairment associated with chemotherapy induced peripheral neuropathy.

DETAILED DESCRIPTION:
Taxanes, a type of chemotherapeutic agent prescribed to breast cancer patients, have a known physical side effect of chemotherapy induced peripheral neuropathy (CIPN). The purpose of this qualitative study is to understand the experience and physical functional side effects of taxanes. This is the first of a two phase study. The overall goal is to identify existing objective physical performance measures to assess functional side effects of taxanes.

ELIGIBILITY:
Inclusion Criteria:

* Women 21-70 years old (Women over 70 are offered chemotherapy less frequently because of their risk benefit ratio. Including them would be a selection bias because of their differential underexposure).
* Initiated taxane-based chemotherapy in the neoadjuvant, adjuvant, or previously untreated metastatic setting.
* The range of exposure to taxane-based chemotherapy will include women on active treatment having received two cycles, to women who are within three months of their last infusion.
* Documented symptoms of CIPN per CTCAE grading criteria (half of sample) or NO symptoms (half of sample) Grade 0 = no CIPN symptoms Grade 1 = mild symptoms Grade 2 = moderate symptoms - prescribed Gabapentin (Neurontin) Grade 3&4= severe symptoms - treated with Gabapentin (Neurontin), treatment plan altered

Exclusion Criteria:

* Physical disabilities - defined by use of assistive devices to complete functional tasks (wheelchair, crutches, prosthetic limbs) prior to starting chemotherapy.
* Current exposure to neurotoxic agents (Navelbine, platinums or other taxanes)
* Pregnancy during chemotherapy treatment
* Diabetes - diagnosed 3 or more years , or insulin dependent, or with clinically established neuropathy
* Previous exposure to chemotherapy or radiotherapy
* HIV positive (high risk for neuropathy)
* Other neurological diseases, such as Multiple Sclerosis
* Other pre-existing neuropathy

Ages: 21 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The semi-structured interviews will be conducted with breast cancer patients of the Rena Rowan Breast Center of the Abramson Cancer Center of the University of Pennsylvania. A purposive sampling strategy in which study participants are recruited based on a particular characteristic of experience of interest, will be used to select breast cancer patients (N=30). Participants will be recruitedwith the goal of having a balanced sample of women who experience documented CIPN (per Common Toxicity Criteria for Adverse Events CTCAE - grading criteria, details below) and those who received a taxane but did not have documented CIPN.
Sampling Method: Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2010-06; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Number of interviews | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Angela DeMichele, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States